CLINICAL TRIAL: NCT02838446
Title: Cognitive Therapy Model: Graded Motor Imagery
Brief Title: Effectiveness of Graded Motor Imagery to Improve Hand Function in Patients With Distal Radius Fracture
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Burcu Dilek, PT, Ass. Prof. Dr., Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 14/06
Record Dates: First submitted 2016-07-11; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Distal Radius Fracture; Pain
MeSH Terms: conditions — Wrist Fractures; Pain | interventions — Cognitive Behavioral Therapy; Rehabilitation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Cognitive Therapy (Experimental): Graded motor imagery program was applied in only intervention group for 8 weeks.
  Interventions: Procedure: Cognitive Therapy
- Control (Active Comparator): Rehabilitation program applied in both groups for 8 weeks. Frequency of the treatment was 2 days in per week and its duration was approximately one hour in one session.
  Interventions: Procedure: Cognitive Therapy

INTERVENTIONS:
Procedure: Cognitive Therapy — Graded Motor Imagery has three stages:
  Lateralisation (2 or 3 weeks) Motor Imagery (2 or 3 weeks) Mirror Therapy (2 or 3 weeks)
  Other Names: Rehabilitation

SUMMARY:
The purpose of this study was to investigate of the effectiveness of Graded Motor Imagery (GMI) on hand functionality in patients with Distal Radius Fracture (DRFx). This study was carried out on 36 patients. These patients were randomly assigned to two groups: classic treatment group (n=19) and GMI group (n=17). Both groups received a 8-week (2 days a week) physical therapy and rehabilitation intervention. Outcome measurements were based on upper extremity functional status (Disability of the Arm Shoulder Hand and Michigan Hand Questionnaire scores), pain (on the rest and during the activity with Visual Analog Scale), range of motion (wrist flexion, extension, ulnar/radial deviation, supination and pronation with goniometer), grip strength (standard grip strength with Jamar hydraulic hand dynamometer; lateral, palmar and pinch strength with pinch meter).

ELIGIBILITY:
Inclusion Criteria:

* ages between 18-65 years
* diagnosed with DRFx which is extra-articular
* managed with pins, internal fixation and/or cast

Exclusion Criteria:

* unwilling or unable to participate
* intra-articular and instable fractures containing other part of the fractures
* fractures related with the malignancy and other neurologic diseases
* existing inflammatory joint condition,
* lack of cognitive function.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Physical Function and Symptoms | 8 weeks
  Disability of the Arm, Shoulder and Hand (DASH) questionnaire scores range from 0 to 100 with a higher score indicating higher degree of disability.

SECONDARY OUTCOMES:
Pain intensity | 8 weeks
  Visual Analog Scale (VAS) is used to evaluate pain intensity. The scale was consisted of a standard line labeled 0 on the left and 10 on the right. (0: no pain, 10: the worst pain).
Normal range of motion | 8 weeks
  Active range of motions of wrist regarding flexion, extension, ulnar deviation, radial deviation, supination and pronation were evaluated with universal goniometer and recorded as degree.
Grip Strength | 8 weeks
  Grip strength was measured in kilograms using a calibrated Jamar Hydraulic Hand Dynamometer with the elbow flexed to 90 degree.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)